CLINICAL TRIAL: NCT02079467
Title: Unrestricted Rehabilitation Following Primary Total Hip Arthroplasty: Implications for Patient Satisfaction and Functional Performance
Brief Title: Unrestricted Rehabilitation Following Primary THA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Veronica Wadey, Staff surgeon, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Miller-01
Record Dates: First submitted 2013-12-04; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis, Hip
Keywords: Arthroplasty, Hip; Replacement, Hip; Postoperative Care; Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard rehabilitation (Active Comparator): Patients randomized to the control group will be managed with "hip precautions" immediately following surgery. They will weight bear on the operative joint as tolerated after surgery. They will be managed as per usual protocol post total hip arthroplasty. They will be transferred from the operative table with an abduction pillow between their legs and will be asked to keep this pillow between their legs while resting in bed and during sleep throughout their course in hospital. During physiotherapy treatments they will not flex the operative hip beyond 90 degrees, internally or externally rotate the operative hip more than 45 degrees, or actively adduct the operative hip past neutral.
  Interventions: Procedure: Standard rehabilitation
- Unrestricted rehabilitation (Experimental): Patients randomized to the treatment group will have no restrictions in their post-operative rehabilitation. They will weight bear on the operative joint as tolerated after surgery. They will be asked to participate in activity as their level of comfort permits and will have no positional restrictions while in bed or completing activities of daily living.
  Interventions: Procedure: Unrestricted rehabilitation

INTERVENTIONS:
Procedure: Unrestricted rehabilitation — Standard care range of motion restrictions will not be used
  Arms: Unrestricted rehabilitation
Procedure: Standard rehabilitation — Standard care range of motion restrictions will remain in place
  Arms: Standard rehabilitation

SUMMARY:
The purpose of this study is to determine whether the form of rehabilitation following primary total hip arthroplasty has an influence on patient satisfaction or functional performance in the eighteen weeks following surgery.

DETAILED DESCRIPTION:
The current standard of care following total hip replacement is to restrict patient activity and range-of-motion with the goal of avoiding dislocation of the operative hip. These restrictions are commonly referred to as "hip precautions". Several recent studies have demonstrated these precautions may be safely abandoned with no increased risk of dislocation when the surgery is carried through an anterior/lateral approach. Previous work has failed to address the issue of patient satisfaction and functional performance when patients are managed with an unrestricted rehabilitation protocol post-operatively. We propose a prospective, randomized clinical trial to determine whether an unrestricted postoperative rehabilitation protocol has an impact on patient satisfaction and functional performance following primary total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 50 years
* Undergoing primary total hip arthroplasty at Holland Orthopaedic and Arthritic Centre

Exclusion Criteria:

* Any previous surgery about the ipsilateral hip
* Patients being considered for simultaneous bilateral total hip arthroplasty
* Patients with a neuromuscular disorder or recognized hypermobility syndrome
* Patients without sufficient language skills to communicate in spoken and written English

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | Six weeks post-operatively
  The test involves measuring the duration of time required for a patient to rise from a standard arm chair, walk 3 metres, turn, walk back to the chair, and sit down.

SECONDARY OUTCOMES:
4-Item Pain Intensity Measure (P4) | Baseline
  The measure involves patients recording the subjective experience of their pain on a scale from 0 - 10 at different times during the day (morning, afternoon, evening) as well as with activity.
Lower extremity functional scale (LEFS) | Baseline
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention.
PROMIS Bank v2.0 - Satisfaction with Social Roles and Activities - Computerized Adaptive Testing | Baseline
  This is a tool developed by the National Institutes of Health (NIH) which uses item response theory to select questions from a validated item bank to get a precise measurement of patient status in a chosen domain.
Timed Up and Go (TUG) | Baseline
  The test involves measuring the duration of time required for a patient to rise from a standard arm chair, walk 3 metres, turn, walk back to the chair, and sit down.
Timed Up and Go (TUG) | Date of discharge following surgery (2 to 6 days post-op, but could be up to 2 weeks)
  The test involves measuring the duration of time required for a patient to rise from a standard arm chair, walk 3 metres, turn, walk back to the chair, and sit down.
Timed Up and Go (TUG) | Eighteen weeks post-operatively
  The test involves measuring the duration of time required for a patient to rise from a standard arm chair, walk 3 metres, turn, walk back to the chair, and sit down.
Six Minute Walk Test (6MWT) | Baseline
  This test involves the measurement of the total distance an individual is able to walk over a period of six minutes along a marked pathway with time allowed to rest as required.
Six Minute Walk Test (6MWT) | Six weeks post-operatively
  This test involves the measurement of the total distance an individual is able to walk over a period of six minutes along a marked pathway with time allowed to rest as required.
Six Minute Walk Test (6MWT) | Eighteen weeks post-operatively
  This test involves the measurement of the total distance an individual is able to walk over a period of six minutes along a marked pathway with time allowed to rest as required.
4-Item Pain Intensity Measure (P4) | Date of discharge following surgery (2 to 6 days post-op, but could be up to 2 weeks)
  The measure involves patients recording the subjective experience of their pain on a scale from 0 - 10 at different times during the day (morning, afternoon, evening) as well as with activity.
4-Item Pain Intensity Measure (P4) | Six weeks post-operatively
  The measure involves patients recording the subjective experience of their pain on a scale from 0 - 10 at different times during the day (morning, afternoon, evening) as well as with activity.
4-Item Pain Intensity Measure (P4) | Eighteen weeks post-operatively
  The measure involves patients recording the subjective experience of their pain on a scale from 0 - 10 at different times during the day (morning, afternoon, evening) as well as with activity.
Lower extremity functional scale (LEFS) | Six weeks post-operatively
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention.
Lower extremity functional scale (LEFS) | Eighteen weeks post-operatively
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention.
PROMIS Bank v2.0 - Satisfaction with Social Roles and Activities - Computerized Adaptive Testing | Six weeks post-operatively
  This is a tool developed by the National Institutes of Health (NIH) which uses item response theory to select questions from a validated item bank to get a precise measurement of patient status in a chosen domain.
PROMIS Bank v2.0 - Satisfaction with Social Roles and Activities - Computerized Adaptive Testing | Eighteen weeks post-operatively
  This is a tool developed by the National Institutes of Health (NIH) which uses item response theory to select questions from a validated item bank to get a precise measurement of patient status in a chosen domain.

CONTACTS AND LOCATIONS:
Overall Officials: Hans J Kreder, MD MPH FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto; Richard Jenkinson, MD MSC FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto; Veronica MR Wadey, BPHE BEd MD MA FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Holland Orthopaedic and Arthritic Centre, Toronto, Ontario, Canada